CLINICAL TRIAL: NCT06457126
Title: Applying the Metacognitive Model to Post-Stroke Emotionalism: A Multiphasic Case Series Piloting the Attention Training Technique
Brief Title: Piloting the Attention Training Technique for Post-Stroke Emotionalism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 333045
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Emotionality; Pseudobulbar Affect; Lability Emotional; Crying
Keywords: Stroke; Post Stroke Emotionalism; Attention Training Technique; Crying Symptoms
MeSH Terms: conditions — Stroke; Crying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Attention Training Technique (Experimental): An audio-recorded 12-minute version will be used and administered with permission and training from the creator of the Attention Training Technique (Professor Adrian Wells). At least four to eight sessions will be administered, given the minimally effective dose is four. Administration will continue until stable effects in the data are observed.
  Interventions: Behavioral: Attention Training Technique

INTERVENTIONS:
Behavioral: Attention Training Technique — Phase 1: Non-concurrent multiple baseline design A-B design where the ATT (B) is introduced sequentially across participants. ATT and baseline (A) will be alternated on a weekly basis.
  Phase 2: Alternating treatment design where an active (B) and passive (C) version of the ATT are rapidly and frequently alternative within the same participant on a weekly basis (e.g., A-B-A-C-A or A-C-A-B-A).
  Other Names: ATT

SUMMARY:
The aim of this mutli-phasic systematic case series is to explore if the Attention Training Technique (ATT) can improve symptoms of Post Stroke Emotionalism. It will teach the ATT to at least three people who have had a stroke at least six months ago, have PSE and are currently receiving support from a Community Neurorehabilitation service in the North West of England. Stroke survivors will also require the support of a carer/loved to record their symptoms on a daily basis. Stroke survivors will attend weekly appointments either at the community service site or via video-call for up to 15 weeks. There is also the option to complete an interview to discuss their experiences of learning the ATT. This study hopes to be the first step in establishing evidence in support of a novel psychological intervention to help improve PSE symptoms.

Phase 1 of the study aims to explore the effects associated with the ATT on PSE symptoms. The primary research questions are:

1a. Is the ATT associated with an improvement of PSE symptoms?

1b. Does this replicate across individual cases?

If these are not initially supported, the ATT delivery will be extended, addressing:

1. c. Is the ATT associated with an improvement of PSE symptoms when some parameters (e.g., frequency and dose) are modified?

   Only if a clear association between ATT and symptom change is demonstrated, will Phase 2 begin.

   Phase 2 aims to understand the relative mechanisms underlying any treatment effect. The primary research question for Phase 2 is:
2. a. Is the ATT associated with a greater change in PSE symptoms than a comparator passive listening intervention (controlling for non-specific factors, (e.g., provision of a credible intervention, task practice and therapist involvement))?

The comparator intervention will be a passive version of the ATT whereby participants are instructed to not follow the instructions on the audio-recording.

Secondary research questions throughout Phase 1 and 2 will address:

1. Is the active ATT (and passive ATT) associated with an improvement in executive functioning, attention, mood and quality of life and is there any difference between the two interventions?

DETAILED DESCRIPTION:
This study is a multi-phasic systematic case series piloting the ATT with stroke survivors presenting with PSE across two phases with extended baselines (A). Phase 1 will utilise a non-concurrent multiple baseline AB design where the ATT (B) is introduced sequentially across participants. Phase 2 will utilise an alternating treatment design where the ATT is compared to a passive listening task (C). To do this, each intervention will be rapidly and frequently alternated within the same participant (ABACA or ACABA). Participants in Phase 2 will be randomised to a predetermined treatment block over a time-limited period; the length of which will be informed by findings in Phase 1.

Sample and Recruitment:

Participants will be stroke survivors who are presenting with PSE and an allocated carer/loved one to support each stroke survivor. As differentiating between PSE and adjustment- distress is difficult during the acute phases of recovery, this study will only recruit people who are at least six months post-stroke.

Stroke survivor participants will be recruited from post-acute community stroke services. Participants will be identified by stroke clinicians during routine clinical practice. They will share this information to service-users and their carers who meet the inclusion criteria as part of their routine care. A Consent to Contact form and Eligibility Form will be completed by the clinician where participants and their carers consent to be contacted by a member of the research team. Those who provide permission to be contacted and are identified by the clinical care team as eligible for screening will be contacted in-person or by email, telephone, or video-call (according to their preference). The initial contact will provide further information about the study, answer any questions and to arrange a screening appointment if they wish to proceed.

Eligibility Screening:

A screening appointment will be organised with interested participants. This will include administration of two screening measures: the TEARS-Q and FAST to determine stroke survivor eligibility for participation. The data obtained initially from these measures will be to ascertain eligibility and not form part of the research data set. If eligible, participants and their carer will be provided with an accessible Participant Information Sheet to enable them to make an informed decision about participation. Follow-up contact will be made one week after the screening appointment, if no response has been received, to provide an opportunity to answer any questions, provide further information about what is entailed and to allow the service-user time to consider whether they would like to take part. If the service-user decides to take part, an initial appointment will be made to take written informed consent using the Consent Form, further explain the protocol for participation and to start the collection of baseline data. Throughout the consenting process, consent will be sought to use the screening measure data as part of the research dataset.

Extended Baseline - Phase 1 and 2:

In the first appointment, participants will be reminded of the study protocol and that the intervention(s) are individual techniques that do not equate to formal therapy. Risk-assessments and distress-management plans will be in place to support participants if they are needed. Participants and their carer will be shown how to complete the PSE primary outcome measures (the daily diaries). Compensatory strategies (e.g., reminders or alarms) will be discussed and tailored to the participants' needs, if required. Pre-intervention measures will be administered. These include: OCS; HADS and WHOQOL-BREF. Relevant demographic information of each participant will be collected using a bespoke demographic questionnaire. This will include data about their age, gender, marital status, nature of their stroke, physical and mental health and medical etc. Subsequent weekly contact will not provide any therapeutic instruction and only collect the daily diary measure data from the participant and their carer. This will continue until stable trends in PSE symptoms are observed for at least three data points.

Intervention:

Phase 1 - The first session will present the participant with a rationale for using the ATT to manage PSE. The pre- intervention credibility questionnaire will be administered. An audio-recorded version of the ATT will then be introduced. Daily diary measure data will be collected from the participant and their carer. Subsequent weekly sessions will include further practice of the ATT and the collection of the daily diary measure data. At least four to eight sessions of the ATT will be administered given the minimally effective dose is four (Heitland et al., 2020). This will continue until stable effects in the data are observed.

Phase 2 - A randomisation procedure will allocate each participant to a predetermined treatment sequence to ascertain which intervention they start with. The first intervention session will provide the participant with a rationale for using either the active ATT (follow the instructions) or passive ATT (do not follow the instructions). The order of the interventions will be randomised and counterbalanced across participants. The pre-intervention credibility questionnaire will be administered. Participants will then be taught both interventions using audio recordings of each in subsequent sessions. The daily diary measure data will be collected at each contact. At the end of predetermined study sequence, participants will be asked about their experience of each intervention and their preferences.

Post-Intervention measures will then be administered in both Phase 1 and 2 in the final intervention session. Again, these include: OCS; HADS and WHOQOL-BREF. The TEARS-Q will also be repeated at this point to ascertain whether there has been any change in their PSE symptoms. The post-intervention credibility questionnaire will also be administered in the last intervention session.

Post-Intervention Interview - Phase 1 and 2:

This will be an optional brief semi-structured interview exploring participants' reaction to/views on the ATT intervention (e.g., what they found helpful and/or unhelpful). This will only take place after the participant has completed their final intervention session.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary clinical diagnosis of an ischemic or haemorrhagic stroke.
* At least six months or more post-stroke
* Reported/observed difficulties with symptoms of PSE (episodes of uncontrollable and unpredictable crying that is not mood congruent and happens in situations that the person would not have otherwise cried)
* Scores between 6-16 on the Testing Emotionalism after Stroke Questionnaire (TEARS-Q; Broomfield et al., 2021)
* Scores > 25 on the Frenchay Aphasia Screening Test (FAST; Enderby, Wood, and Wade 1987).
* Aged 18 or over.
* Has the Mental Capacity (Mental Capacity Act, 2005) to provide informed consent.
* Has carer support and consents to their carer being involved.
* Proficient in English Language
* No anticipated changes to antidepressant medication (if applicable).

Exclusion Criteria:

* Less than six months post-stroke
* Presenting with PSE without a primary diagnosis of an ischemic or haemorrhagic stroke and/or as a result of another neurological condition.
* Hyper acutely or acutely unwell with concurrent medical conditions.
* Receiving palliative or end of life care.
* Severe or distressing behaviours that may impede on engagement or cause further distress.
* Visual or hearing impairment unable to be corrected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-06-24 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Daily Diaries - Stroke Survivor and Carer | Baseline: daily from time one to end of baseline. Intervention: daily from intervention time point one to end of intervention period (minimum of four to eight weeks to maximum of 15-weeks post-baseline).
  A repeatable observational measure of PSE symptom frequency and uncontrollability. A repeatable observational measure of PSE symptom frequency and uncontrollability did not exist during the development of the study. It is typical in SCEDs for clinicians to develop measures such as these (Krasny-Pacini and Evans, 2018). A participant diary has been developed in addition to a carer diary to enable measurement of inter-rater reliability. In recognition that PSE symptoms may present on a continuum of tearfulness through to uncontrollable sobbing, a Likert scale has been developed within the measure to ascertain the severity of presenting symptoms.
  This will measure:
  1. Time of sudden onset tearfulness or crying
  2. How tearful or how much the person cried
  3. Whether the tearfulness or crying was expected or unexpected.
  4. Emotions associated with start of tearfulness or crying.
  5. Visual analogue scale measure of uncontrollability to controllability.

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HADS) | Baseline time one; Post-intervention (a minimum of four to eight weeks to a maximum of 15-weeks from end of baseline).
  An objective measure of anxiety and depression validated for use in stroke (Zigmond and Snaith, 1983; Sagen Vik, Finset, Moum, Vik and Dammen, 2022). It has 14-items rated on a scale from 0-3. Anxiety (7 items; maximum score 21) and Depression (7 items; maximum score 21). In response to each item, participants must select the response most appropriate to how they have felt over the past week. Higher scores indicate a worse outcome (e.g., scores between 11 and 21 indicate clinical levels of anxiety or depression).
The Oxford Cognitive Screen (OCS) | Baseline time one; Post-intervention (a minimum of four to eight weeks to a maximum of 15-weeks from end of baseline).
  A recommended brief cognitive assessment for stroke (Quinn, Elliott, and Langhorne, 2018). Includes ten tasks assessing executive function, attention, language, memory, number processing and praxis (Demeyere et al., 2016; Demeyere et al., 2015). The OCS will also be used as a descriptive tool for the cognitive profile of the sample.
  Naming (max score 4) Semantics (3) Orientation (4) Visual Field (4) Sentence Reading (15) Number Writing (3) Calculation (4) Hearts (50) Space Asymmetry (less than -2 = right egocentric neglect. more than 3 = left neglect) Object Asymmetry (ess than -1 = right allocentric neglect. more than = left neglect) Imitation (12) Verbal Recall / Recognition (4) Episodic Recognition (4) Executive Score (-1)
  Lower scores indicate greater cognitive impairment with the exception of the executive score and asymmetry tests. Higher executive score indicates greater cognitive impairment. Asymmetry scores are as above.
World Health Organisation Quality of Life Scale (WHOQOL-BREF) | Baseline time one; Post-intervention (a minimum of four to eight weeks to a maximum of 15-weeks from end of baseline).
  A shorter, easier to administer version of the WHO-QOL and has been validated for use in stroke (Martini, Ningrum, Abdul-Mumin and Yi-Li, 2022). It is a 26-item self-report questionnaire measuring physical, psychosocial, and environmental QoL, overall QoL and health - based on the last two weeks. Raw scores are rated between 1 and 5. Maximum transformed score = 100. Higher scores indicate higher quality of life.
Focus of Attention Rating Scale | Weekly during intervention (across a minimum of four to eight weeks to a maximum of 15-weeks).
  This will be used as a manipulation check to ascertain if the ATT is working as it aims to. It includes a 7-point rating scale to measure the change from an internal to external focus of attention (Wells, 2009). Lower scores indicate an external focus of attention. Higher scores indicate an internal focus of attention.
The Testing Emotionalism after Recent Stroke Questionnaire (TEARS-Q) | Screening appointment and post-intervention (ie., a minimum of four to eight weeks to a maximum of 15-weeks from end of baseline).
  A self-report questionnaire to identify stroke survivors experiencing sudden onset crying. It has been psychometrically validated (Broomfield et al., 2021). Maximum score = 16. Higher scores indicate higher probability of post stroke emotionalism.

OTHER OUTCOMES:
Post-Intervention Interview | 1-week following the end of intervention (ie., a minimum of five to nine weeks to a maximum of 15-weeks post-baseline dependent on the length of the intervention according to participant needs).
  An optional brief semi-structured interview exploring participants' reaction to/views on the ATT intervention (e.g., what they found helpful and/or unhelpful).

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wells, Study Director — University of Manchester
Locations (2):
- United Kingdom (2):
  - Manchester University NHS Foundation Trust, Manchester
  - Northern Care Alliance, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow, D., Nock, M., & Hersen, M. (2009) Single Case Experimental Design: Strategies for Studying Behaviour Change (3rd ed.) Pearson.
- [Background] Broomfield NM, West R, House A, Munyombwe T, Barber M, Gracey F, Gillespie DC, Walters M. Psychometric evaluation of a newly developed measure of emotionalism after stroke (TEARS-Q). Clin Rehabil. 2021 Jun;35(6):894-903. doi: 10.1177/0269215520981727. Epub 2020 Dec 21. PMID 33345598
- [Background] Broomfield NM, West R, Barber M, Quinn TJ, Gillespie D, Walters M, House A. TEARS: a longitudinal investigation of the prevalence, psychological associations and trajectory of poststroke emotionalism. J Neurol Neurosurg Psychiatry. 2022 Apr 28:jnnp-2022-329042. doi: 10.1136/jnnp-2022-329042. Online ahead of print. PMID 35483914
- [Background] Fitzgerald S, Gracey F, Broomfield N. Post-stroke emotionalism (PSE): a qualitative longitudinal study exploring individuals' experience with PSE. Disabil Rehabil. 2022 Dec;44(25):7891-7903. doi: 10.1080/09638288.2021.2002439. Epub 2021 Nov 16. PMID 34784814
- [Background] Fitzgerald S, Gracey F, Trigg E, Broomfield N. Predictors and correlates of emotionalism across acquired and progressive neurological conditions: A systematic review. Neuropsychol Rehabil. 2023 Jun;33(5):945-987. doi: 10.1080/09602011.2022.2052326. Epub 2022 Mar 24. PMID 35323084
- [Background] Gillespie DC, Cadden AP, West RM, Broomfield NM. Non-pharmacological interventions for post-stroke emotionalism (PSE) within inpatient stroke settings: a theory of planned behavior survey. Top Stroke Rehabil. 2020 Jan;27(1):15-24. doi: 10.1080/10749357.2019.1654241. Epub 2019 Aug 28. PMID 31461389
- [Background] Gillespie DC, Halai AD, West RM, Dickie DA, Walters M, Broomfield NM. Demographic, clinical and neuroimaging markers of post-stroke emotionalism: A preliminary investigation. J Neurol Sci. 2022 May 15;436:120229. doi: 10.1016/j.jns.2022.120229. Epub 2022 Mar 21. PMID 35378397
- [Background] Knowles MM, Foden P, El-Deredy W, Wells A. A Systematic Review of Efficacy of the Attention Training Technique in Clinical and Nonclinical Samples. J Clin Psychol. 2016 Oct;72(10):999-1025. doi: 10.1002/jclp.22312. Epub 2016 Apr 29. PMID 27129094
- [Background] McAleese N, Guzman A, O'Rourke SJ, Gillespie DC. Post-stroke emotionalism: a qualitative investigation. Disabil Rehabil. 2021 Jan;43(2):192-200. doi: 10.1080/09638288.2019.1620876. Epub 2019 May 28. PMID 31136206
- [Background] Wells, A. (1990). Panic disorder in association with relaxation induced anxiety: An attentional training approach to treatment. Behavior therapy, 21(3), 273-280. https://doi.org/10.1016/S0005-7894(05)80330-2
- [Background] Wells A. Breaking the Cybernetic Code: Understanding and Treating the Human Metacognitive Control System to Enhance Mental Health. Front Psychol. 2019 Dec 12;10:2621. doi: 10.3389/fpsyg.2019.02621. eCollection 2019. PMID 31920769